CLINICAL TRIAL: NCT06269900
Title: Dexamethasone for Treating Severe Hospital-acquired Pneumonia in Critically Ill Patients With a Proinflammatory Phenotype, an International Phase III, Double-blind, Placebo-controlled, Randomized Trial
Brief Title: Dexamethasone for Treating Severe Hospital-acquired Pneumonia in Critically Ill Patients With a Proinflammatory Phenotype
Acronym: HAP-DEX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC23_0358
Record Dates: First submitted 2024-02-05; First posted 2024-02-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hospital Acquired Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexamethasone + standard of care (Experimental): * Dexamethasone 0.2mg.kg-1.day-1 intravenous for a minimal duration of 5 days, and a maximal duration of 7 days in case of persistence of ARDS criteria (PaO2/FiO2 ratio < 300).
  * Standard of care: antimicrobial therapy in compliance with European guidelines. Briefly, intravenous antimicrobial therapy with the narrowest spectrum to cover at-risk and/or identified pathogens for 7-8 days.
  Interventions: Drug: Dexamethasone
- Placebo + Standard of care (Placebo Comparator): * Placebo 0.2mg.kg-1.day-1 intravenous for 5 days and a maximal duration of 7 days in case of persistence of ARDS criteria (PaO2/FiO2 ratio < 300).
  * Standard of care: antimicrobial therapy in compliance with European guidelines. Briefly, intravenous antimicrobial therapy with the narrowest spectrum to cover at-risk and/or identified pathogens for 7-8 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone phosphate injection is given as a slow injection or infusion (intravenous drip) into the veins.
  Arms: dexamethasone + standard of care
Drug: Placebo — Placebo injection is given as a slow injection or infusion (intravenous drip) into the veins.
  Arms: Placebo + Standard of care

SUMMARY:
Determine the efficacy of dexamethasone plus standard of care (SOC) as compared to placebo plus SOC for treating severe hospital-acquired pneumonia in critically ill patients with a proinflammatory phenotype; It's an international phase III, double-blind, placebo-controlled, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Hospital-acquired pneumonia (HAP) according to European guidelines (Torres et al. Eur Respir J 2017): Association of two criteria among (body temperature > 38°C, leukocytosis>12000 cells per mL, leucopenia <4000 cells per mL and purulent pulmonary secretions), appearance of a new infiltrate or change in an existing infiltrate on chest radiography, and respiratory sample (Sputum, AET, BAL, mini-BAL or blind BAL) collected for bacteriological diagnosis (results can be pending at inclusion). The diagnosis of HAP can have been made outside of ICU. Diagnosis is done at least 48 hours after hospital admission.
* HAP severity defined as a PaO2/FiO2 ratio < 300 under mechanical ventilation.
* Biological systemic inflammatory response defined as CPR≥ 150 mg/L (15 mg/dL)*
* Receiving curative antimicrobial therapy for the current episode of HAP pneumonia for less than 48 hours.
* Informed consent from a legal representative, or emergency procedure (when possible, according to national regulation, see below). If it is not possible to obtain the patient consent prior the inclusion (comatose patients), patient consent for the study continuation will be obtained as soon as deemed possible.
* Person insured under a health insurance scheme.
* Female of childbearing age who agree and who are able to comply with effective contraception for the 28 first days of the study.

Exclusion Criteria:

* Pregnant women (serum or urine test), breastfeeding women.
* Patient under legal protection (incl. under guardianship or trusteeship).
* Hypersensitivity to dexamethasone and hypersensitivity to all of its excipients
* Ongoing administration of glucocorticoid at the time of randomisation, such as for COVID-19 infection requiring supplemental oxygen therapy
* Severe septic shock (norepinephrine > 0.4 microg/kg/min and serum lactate level greater than 2 mmol/L) at the time of randomisation
* Prolonged use of corticosteroids at a mean minimum dose of 0.3 mg/kg/day of prednisone equivalent for >3 weeks in the past 60 days
* Uncontrolled viral (hepatitis,herpes, zona, varicella) or systemic fungal infection
* Immunosuppression pre-existing to hospitalisation (severe lymphopenia < 500 lymphocytes/mm3, hematologic cancer, aplasia, chemotherapy/radiotherapy for cancer within 3 months prior to the inclusion, or anti-graft rejection drug).
* Uncontrolled psychotic disorder (acute or chronical)
* Patients not expected to survive for more than 48 hours.
* Participation in another drug clinical trial :

  * testing steroids or anti-graft rejection drug or chemotherapy- radiotherapy for cancer
  * And / Or testing a drug regimen with a known interaction with dexamethasone,
  * And / Or whose implementation would alter the HAP-DEX 6-month follow-up, notably the collection of the primary outcome.
  * Situations that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate at the test-of-cure visit (TOC visit) | Day 8-10
  It's a hierarchic procedure. First, we will test the dexamethasone superiority on the clinical cure rate at the test-of-cure visit realized 8 days (acceptable time frame Day 8-10) after randomization or at the ICU discharge (if it occurs before).
The rate of all-cause mortality on Day 28. | Day 28

SECONDARY OUTCOMES:
Rate of death | Month 3 , Month 6
  All-cause mortality
Rate of pleural empyema at Day 28. | Day 28
Rate of microbiological failure | Toc 1 day visit
Rate of pneumonia relapse | day 28
Duration of hospitalization and hospital-free days | Month 6
Rates of non-respiratory hospital-acquired infection | Day 28
Antibiotic-free days at Day 28 | Day 28
Duration of invasive mechanical ventilation and invasive mechanical ventilation-free days | Month 6
Rate of SUSAR ( suspected unexpected serious adverse reaction) and AE ( Adverse event) | day 28
  * Rate of serious adverse reactions and suspected unexpected serious adverse reaction (SUSAR)
  * Rate of metabolic adverse events
Rate of gastric ulcer | day 28
Anxiety and depression were measured with the HADS (Hospital Anxiety and Depression Scale | month 3, month 6
  Changes in anxiety and depression were measured with the HADS (Hospital Anxiety and Depression Scale ) scale in order to assess the acceptability of dexamethasone from the patients' perspectives
Changes in subjective well-being with the Satisfaction With Life Scale (SWLS) | month 3, month 6
  Changes in subjective well-being from M3 to M6 measured with the Satisfaction With Life Scale (SWLS) in order to assess the acceptability of dexamethasone from the patients' perspectives
Changes in health-related quality of life measured with the Short Form (SF)-36 | month 3, month 6
  Changes in health-related quality of life with the Short Form (SF)-36 scale in order to assess the acceptability of dexamethasone from the patients' perspectives:
the cost-effectiveness analysis (CEA ) will estimate an incremental cost-effectiveness ratio (ICER) | month 6
  We will assess the economic efficiency of dexamethasone plus standard of care compared to standard of care by performing a cost-effectiveness analysis (CEA) using QALYs (Quality-Adjusted Life-Years) as a measure of health outcomes. the CEA will estimate an incremental cost effectiveness ratio (ICER) using a collective perspective; The ICER will be expressed in terms of costs per QALY gained.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ROQUILLY, Principal Investigator — Nantes University Hospital
Locations (21):
- France (21):
  - Chu Amiens, Amiens
  - CHU Angers, Angers
  - Chu Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CHU Clermont - Ferrand, Clermont-Ferrand
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Beaujon, Clichy
  - CHU Raymond Poincaré, Garches
  - Chu Grenoble, Grenoble
  - CHU Limoges, Limoges
  - CHU Marseille, Marseille
  - Chu Nancy, Nancy
  - CHU Nantes (HGRL), Nantes
  - CHU Nantes, Nantes
  - Chu Nimes, Nîmes
  - CHU Pitié Salpétrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided